CLINICAL TRIAL: NCT01801072
Title: Seizure Prophylaxis in Aneurysm Repair
Acronym: SPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Aditya S. Pandey, MD, Professor of Neurosurgery, Chair, Department of Neurosurgery, Professor of Radiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00064523
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Aneurysms; Seizure
MeSH Terms: conditions — Intracranial Aneurysm; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levetiracetam (Active Comparator): 500 mg intravenous dose during the operative case then 500 mg orally twice a day for a total of seven days.
  Interventions: Drug: Levetiracetam
- No levetiracetam (No Intervention): No levetiracetam during the operative phase.

INTERVENTIONS:
Drug: Levetiracetam — Details covered in Arm Descriptions.
  Other Names: Keppra
  Arms: Levetiracetam

SUMMARY:
After a thorough review of the existing literature as well as a review of our own practice, the investigators have concluded that the decision to treat patients undergoing aneurysm repair with levetiracetam has reached true clinical equipoise. In other words, the investigators cannot favor a decision to either administer or not administer this drug in these patients based on the existing information. The utility of anti-epileptic prophlaxis in the perioperative period for patients undergoing intracranial aneurysm repair remains a common practice that is not supported by the current literature that includes retrospective analyses as well as prospective trials for similar but not identical types of patients. The investigators propose to settle this dilemma by performing a prospective randomized trial in patients undergoing aneurysm repair in order to definitively determine if the common practice of perioperative antiepileptic drug administration has any utility. The study will be extended to June 2024 to allow for a 5 year follow up of the last enrolled patient in June, 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Presence of intracranial aneurysm (with or without rupture)
* Treating surgeon has recommended surgical repair of the aneurysm

Exclusion Criteria:

* History of seizures within last 10 years
* History of epilepsy
* History of prior stroke
* Currently prescribed medication with anti-epileptic activity (keppra, dilantin, tegretol, lamictal, topamax, etc.)
* Brain tumor
* Pregnant or nursing woman
* Known levetiracetam allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aditya S Pandey, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levetiracetam | No Levetiracetam
Started | 40 | 42
Hospitalization | 35 | 39
Completed | 11 (Subjects that were reached for the five year follow-up phone call.) | 17 (Subjects that were reached for the five year follow-up phone call.)
Not Completed | 29 | 25
Not completed — Lost to Follow-up | 17 | 14
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Death | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | No Levetiracetam | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 34 | 65
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 13 | 12 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Seizure
Description: Incidence of seizure reported as number of participants who had at least one seizure within the relevant date range. Data collected at hospital discharge, 1-2 months, 4-6 months, 6-12 months, and 5 years. Data is not cumulative. Counts reflect the number of participants who experienced a seizure since their previous check-in.
Time Frame: 5 years from procedure
Population: The number of participants analyzed differs from the totals enrolled as some subjects withdrew consent after randomization or were taken out of the study due to physician decision.
Measure: Count of Participants; unit: Participants
Arm/Group | Levetiracetam | No Levetiracetam
Number analyzed (Participants) | 40 | 42
Participants
  Hospitalization: number analyzed (Participants) | 35 | 39
  Hospitalization | 2 | 1
  1-2 Months: number analyzed (Participants) | 29 | 31
  1-2 Months | 0 | 0
  4-6 Months: number analyzed (Participants) | 26 | 27
  4-6 Months | 0 | 0
  6-12 Months: number analyzed (Participants) | 14 | 16
  6-12 Months | 0 | 0
  5 years: number analyzed (Participants) | 10 | 16
  5 years | 1 | 2

2. Secondary Outcome: Duration of Seizure
Description: Duration of seizure
Time Frame: To compare duration of seizure in each randomization group
Population: While this was originally intended to be a measure collected for this study, the unpredictability of seizure occurrences and the consequent challenges with observing them consistently resulted in our being unable to collect this data from participants.
Arm/Group | Levetiracetam | No Levetiracetam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Levetiracetam | No Levetiracetam
All-Cause Mortality (participants affected / at risk) | 7/40 | 8/42
Serious Adverse Events (participants affected / at risk) | 2/40 | 2/42
Other Adverse Events (participants affected / at risk) | 7/40 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=40) | No Levetiracetam (N=42)
Acute Right Vision Loss (Eye disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=40) | No Levetiracetam (N=42)
Unexplained Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Delirium (Nervous system disorders) | 1 | 0
Patient received extra Keppra (Product Issues) | 1 | 0 — Participant was randomized to the Keppra arm. Patient was inadvertently discharged with a 30-day supply of Keppra. Once the study team became aware of this, the patient was fully instructed how to taper off Keppra.
Seizure (Nervous system disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01801072/Prot_SAP_000.pdf